CLINICAL TRIAL: NCT06366958
Title: Arthroscopic Versus Open Excision of Dorsal Wrist Ganglion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelaal Sayed, resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dorsal wrist ganglion
Record Dates: First submitted 2024-01-13; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Hand Ganglion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Other): arthroscopic excision
  Interventions: Procedure: excision of dorsal wrist ganglion
- group 2 (Other): open excision
  Interventions: Procedure: excision of dorsal wrist ganglion

INTERVENTIONS:
Procedure: excision of dorsal wrist ganglion — open and arthroscopic excision of dorsal wrist ganglion

SUMMARY:
compare recurrence rates after open and arthroscopic excision of dorsal wrist ganglion

DETAILED DESCRIPTION:
DORSAL GANGLIONS (DGS) are one of the most frequent problems of the wrist. They represent benign soft tissue tumors that frequently remain asymptomatic. Suggested causes include trauma to the scapholunate joint, degeneration of tissue lining a tendon or sheath near the joint, and synovial herniation in most cases, diagnosis is based on history and physical examination. Patients seek treatment when these ganglions become associated with pain, weakness, interference with activities, and an increase in size Other than observation, nonoperative treatment such as closed rupture, ganglion puncture, and needle aspiration is associated with relatively higher rates of recurrenceas high as 78%. Surgical treatment with either open or arthroscopic excision is therefore offered with a lower risk of recurrence. Whereas open excision has historically been the traditional method of surgical treatment, arthroscopic excision has been suggested as a potentially more favorable alternative. Proponents of wrist arthroscopy proclaim an advantage of decreased postoperative pain, earlier return of functions, and a smaller incision. Moreover, preliminary and subsequent studies have described arthroscopic DG excision as having equal or lower rates of recurrence. However, the results of arthroscopic versus open procedures have never been directly compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary, simple DG with no underlying pathology of the wrist who sought surgical treatment.

Exclusion Criteria:

* 1. Prior ganglion treatment (rupture, puncture, aspiration, or excision) 2. Previous surgery 3. History of a fracture 4. Ligamentous tear or wrist instability 5. Patients with major medical problems 6. Unacceptable anesthetic risks, 7. Acquired or congenital abnormalities of wrist function or motion

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
comparison of recurrence rate after open versus arthroscopic excision of dorsal wrist ganglion | one year
  compare recurrence rate within one year after intervension

SECONDARY OUTCOMES:
compare post operative pain ,range of motion ,hang grip strength and post operative scar after open versus arthroscopic excision of dorsal wrist ganglion | one year
  compare post operative pain scaled from 1-10 (VAS score) range of wrist motion in degrees ( using goniometer ) hand grip strength in kilograms (using dynamometer)

REFERENCES:
- [Background] Meena S, Gupta A. Dorsal wrist ganglion: Current review of literature. J Clin Orthop Trauma. 2014 Jun;5(2):59-64. doi: 10.1016/j.jcot.2014.01.006. Epub 2014 Jun 3. PMID 25983472 (Retraction: PMID 34589409 J Clin Orthop Trauma. 2020 Sep 17;11(Suppl 5):S916)
- [Background] Konigsberg MW, Tedesco LJ, Mueller JD, Ball JR, Wu CH, Kadiyala RK, Strauch RJ, Rosenwasser MP. Recurrence Rates of Dorsal Wrist Ganglion Cysts After Arthroscopic Versus Open Surgical Excision: A Retrospective Comparison. Hand (N Y). 2023 Jan;18(1):133-138. doi: 10.1177/15589447211003184. Epub 2021 Apr 1. PMID 33789496